CLINICAL TRIAL: NCT00001420
Title: Studies of the Pathogenesis and Natural History of Psoriatic Arthritis
Brief Title: Study of Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950082; 95-AR-0082
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: Lymphocytes; Cytokines; Apoptosis; Psoriasis; Genetics; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

SUMMARY:
This study will examine the genetic and immune factors involved in the cause and development of psoriatic arthritis-a disease of both the skin and joints. It will describe the medical features and natural course of the disease and determine participants' eligibility for experimental treatment protocols.

Patients with known or suspected psoriatic arthritis 5 years of age and older and their relatives may enroll in this study. Patients will be evaluated with a medical history and physical examination, electrocardiogram, blood tests and X-rays. Additional procedures may include:

1. Leukapheresis-Collection of white blood cells for genetic analysis. Whole blood is collected through a needle placed in an arm vein. The blood circulates through a machine that separates it into its components. The plasma is removed and the cells are returned to the body through a second needle placed in the other arm.
2. Skin biopsy-Removal of a small skin sample for microscopic analysis. An area of skin is numbed with an anesthetic and one to three small circular portions (about 1/4 inch in diameter) are cut and removed.
3. Joint aspiration-Removal of a small sample of synovial fluid (lubricating joint fluid). An area of skin around the biopsy site is numbed with an anesthetic, and a needle is inserted into the joint to pull out a small fluid sample.
4. Synovial needle biopsy-Removal of a small sample of synovial tissue (tissue lining the joint). An area of skin around the biopsy site is numbed with an anesthetic and a large needle is inserted into the joint. A smaller needle attached to a syringe is then placed inside the larger needle and small pieces of synovial tissue are removed.
5. Genetic studies-Saliva and blood samples will be collected for gene testing. Saliva is collected by rinsing the mouth with a tablespoon of salt water and spitting into a test tube.

Patients will be followed once or twice a year and may be evaluated for participation in an experimental treatment study.

Participating relatives of patients will fill out a brief medical history questionnaire and provide a DNA sample (blood sample or tissue swab from the inside of the cheek).

DETAILED DESCRIPTION:
Patients with known or suspected psoriatic arthritis will be evaluated at the Clinical Center. Studies will include characterization of the clinical and laboratory features of the disease, research studies of the natural history and pathogenesis, genetic studies, and determination of the patient's eligibility to enter experimental therapeutic protocols. Patients may be asked to contribute blood, skin or synovial membrane samples for immunologic and genetic research studies.

ELIGIBILITY:
INCLUSION CRITERIA:

Psoriatic arthritis (proven or suspected) or;

Family history of psoriasis or psoriatic arthritis (i.e. family members of patients with psoriasis or psoriatic arthritis); and

Willingness and ability of the subject or guardian to give informed consent.

EXCLUSION CRITERIA:

Concomitant medical problems which would confound the interpretation of immunological studies.

Concomitant medical, surgical or other conditions for which inadequate facilities or funds are available to support their care at the NIH.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 999
Dates: Start 1995-03; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker JN. The pathophysiology of psoriasis. Lancet. 1991 Jul 27;338(8761):227-30. doi: 10.1016/0140-6736(91)90357-u. No abstract available. PMID 1676787
- [Background] Espinoza LR, Cuellar ML, Silveira LH. Psoriatic arthritis. Curr Opin Rheumatol. 1992 Aug;4(4):470-8. PMID 1503870
- [Background] Moll JM, Wright V. Psoriatic arthritis. Semin Arthritis Rheum. 1973;3(1):55-78. doi: 10.1016/0049-0172(73)90035-8. No abstract available. PMID 4581554